CLINICAL TRIAL: NCT06740747
Title: Intermittierende Theta-Burst-Stimulation Zur Verbesserung Von Negativsymptomatik Und Kognition Bei Schizophrenie
Brief Title: Intermittent Theta-Burst Stimulation to Improve Negative Symptoms and Cognition in Schizophrenia
Acronym: ITBS-NKS-2024
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Schülke, Rasmus Dr., Principal Investigator, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11473_BO_S_2024
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia Patients
Keywords: iTBS; intermittent theta-burst stimulation; negative symptoms; cognition; schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iTBS (Experimental): Active intermittent theta-burst stimulation of the cerebellar vermis and the left dorsolateral prefrontal cortex
  Interventions: Device: Intermittent theta-burst stimulation
- Sham iTBS (Sham Comparator): Sham intermittent theta-burst stimulation of the cerebellar vermis and the left dorsolateral prefrontal cortex
  Interventions: Device: Sham intermittent theta-burst stimulation

INTERVENTIONS:
Device: Intermittent theta-burst stimulation — Intermittent theta-burst stimulation, applied sequentially to the cerebellar vermis and the left dorsolateral prefrontal cortex
  Arms: iTBS
Device: Sham intermittent theta-burst stimulation — Sham intermittent theta-burst stimulation, applied sequentially to the cerebellar vermis and the left dorsolateral prefrontal cortex
  Arms: Sham iTBS

SUMMARY:
The planned randomized, sham-controlled, double-blind, monocentric study aims to evaluate the effectiveness of intermittent Theta-Burst Stimulation (iTBS) on negative symptoms and cognitive deficits in schizophrenia. Both the cerebellar vermis and the left dorsolateral prefrontal cortex will be stimulated successively within the same session.

The goal of this trial is to learn if intermittent theta-burst stimulation (iTBS) of the cerebellum and the left dorsolateral prefrontal cortext (DLPFC) can treat negative symptoms and improve cognition in patients with schizophrenia. The main question it aims to answer is:

Does iTBS of the cerebellum and the left DLPFC improve negative symptoms in patients with schizophrenia? Researchers will compare iTBS to sham stimulation to see if iTBS improves negative symptoms.

Participants will:

* Receive 10 sessions of iTBS over the course of 2 weeks
* Undergo extensive examination before iTBS treatment, immediately after iTBS treatment and 4 weeks after iTBS treatment. The examination includes assessment of negative symptoms; psychometric assessment of cognition, social cognition, depressive symptoms; functional magnetic resonance imaging; assessment of eye movements; blood and saliva sampling; assessment of adverse events and stimulation associated sensations.

The study thus seeks to determine whether iTBS of the fronto-cerebellar network might improve negative symptoms and cognition by altering the network's functional activity. Additionally, it will investigate whether a pro-inflammatory cytokine profile could affect iTBS outcomes and whether inflammatory markers could be affected by iTBS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (ICD-10: F20.-)
* Age: 18-65 years
* Ability to give informed consent
* Signed informed consent form

Exclusion Criteria:

* Any electronic implants
* Non-MRI-compatible metal implants (e.g., pacemaker, cochlear implant, insulin pump, metal fragment injuries, work in the metal-processing industry)
* Non-TMS-compatible metal implants (compatible items include: earrings, piercings, dental fillings, crowns, implants)
* Claustrophobia
* Epilepsy
* History of traumatic brain injury within the last 3 months
* History of stroke
* Active central nervous system (CNS) infection
* History of CNS infection within the last 3 months
* Pregnancy
* Current drug, medication, or alcohol abuse
* Simultaneous participation in another clinical trial
* Planned changes in psychopharmacological medication within the next 2 weeks
* Severe physical illnesses that could endanger the patient, affect the examinations or make the MRI scanning cause additional burden

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in negative symptoms | From enrollment to the end of iTBS treatment
  Change in negative symptoms, measured with the Clinical Assessment Interview for Negative Symptoms (CAINS). Higher CAINS scores correspond to more negative symptoms. The minimum total score is 0 points, the maximum total score is 52 points.

SECONDARY OUTCOMES:
Change in negative symptoms at 4-week follow-up | From enrollment to follow-up 4 weeks after the end of iTBS treatment
  Change in negative symptoms, measured with the Clinical Assessment Interview for Negative Symptoms (CAINS). Higher CAINS scores correspond to more negative symptoms. The minimum total score is 0 points, the maximum total score is 52 points.
Speech-gesture rating task | From enrollment to the end of iTBS treatment
  Accuracy and speed of evaluations in the Speech-Gesture Rating Task.
Speech-gesture rating task at 4-week follow-up | From enrollment to follow-up 4 weeks after the end of iTBS treatment
  Accuracy and speed of evaluations in the Speech-Gesture Rating Task at 4-week follow-up.
Eye-Tracking Task | From enrollment to the end of iTBS treatment
  Changes in eye movements in the Eye-Tracking Task.
Eye-Tracking Task at 4-week follow-up | From enrollment to 4 weeks after the end of iTBS treatment
  Changes in eye movements in the Eye-Tracking Task at 4-week follow-up.
Reading the Mind in the Eyes Test | From enrollment to 4 weeks after the end of iTBS treatment
  Reading the Mind in the Eyes Test.
Reading the Mind in the Eyes Test at 4-week follow-up | From enrollment to 4 weeks after the end of iTBS treatment
  Reading the Mind in the Eyes Test at 4-week follow-up.
N-Back Test | From enrollment to the end of iTBS treatment
  Working memory performance in the N-Back Test (sensitivity index).
N-Back Test at 4-week follow-up | From enrollment to the end of iTBS treatment
  Working memory performance in the N-Back Test (sensitivity index) 4 weeks after the end of iTBS treatment.
FMRI: Resting-state functional connectivity | From enrollment to the end of iTBS treatment
  Changes in resting-state functional connectivity in functional magnetic resonance imaging. Focus on connectivity between cerebellar vermis and DLPFC.
FMRI: Resting-state functional connectivity at 4-week follow-up | From enrollment to 4 weeks after the end of iTBS treatment
  Changes in resting-state functional connectivity in functional magnetic resonance imaging. Focus on connectivity between cerebellar vermis and DLPFC.
FMRI: Task-related functional connectivity | From enrollment to the end of iTBS treatment
  Changes in task-related functional connectivity in functional magnetic resonance imaging, for the N-Back-task and the speech-gesture rating task.
FMRI: Task-related functional connectivity at 4-week follow-up | From enrollment to 4 weeks after the end of iTBS treatment
  Changes in task-related functional connectivity in functional magnetic resonance imaging, for the N-Back-task and the speech-gesture rating task.
Inflammatory cytokines | From enrollment to the end of iTBS treatment
  Concentrations of inflammatory cytokines (especially IL-6 and TNF-α) in serum and saliva.
Inflammatory cytokines at 4-week follow-up | From enrollment to 4 weeks after the end of iTBS treatment
  Concentrations of inflammatory cytokines (especially IL-6 and TNF-α) in serum and saliva.
Stimulation-associated perceptions | From the beginning of each iTBS stimulation to after the end of each iTBS stimulation
  Stimulation-associated perceptions, measured using the TMS Adverse Events and Associated Sensations Questionnaire (TMSensQ, Section IV), after each iTBS session.
Therapy dropout rate | From the beginning of iTBS treatment to the end of iTBS treatment
  Therapy dropout rate (i.e. study termination).
Serious Adverse Events (SAEs) | From the beginning of iTBS treatment to the end of iTBS treatment
  Serious Adverse Events (SAEs), measured using TMSensQ (Section V).
Self-reported depression: BDI-II | From enrollment to the end of iTBS-treatment
  Self-reported depression, measured using the Beck Depression Inventory-II (BDI-II). Higher scores correspond to more depressive symptoms. The minimum total score is 0 points, the maximum total score is 63 points.
Self-reported depression at 4-week follow-up: BDI-II | From enrollment to 4 weeks after the end of iTBS-treatment
  Self-reported depression, measured using the Beck Depression Inventory-II (BDI-II). Higher scores correspond to more depressive symptoms. The minimum total score is 0 points, the maximum total score is 63 points.
Self-rated gesture perception and production: BAG | From enrollment to the end of iTBS-treatment
  Change in self-rated gesture perception and production, measured using the Brief Assessment of Gestures (BAG) questionnaire. Higher BAG scores correspond to greater engagement with or reliance on gestures in communication and indicate stronger tendencies to produce or perceive gestures effectively in different contexts. The minimum total score is 12 points, the maximum total score is 60 points.
Self-rated gesture perception and production at 4-week follow-up: BAG | From enrollment to 4 weeks after the end of iTBS-treatment
  Change in self-rated gesture perception and production, measured using the Brief Assessment of Gestures (BAG) questionnaire. Higher BAG scores correspond to greater engagement with or reliance on gestures in communication and indicate stronger tendencies to produce or perceive gestures effectively in different contexts. The minimum total score is 12 points, the maximum total score is 60 points.
Epigenetic changes of neurotrophic and immunological factors | From enrollment to the end of iTBS treatment
  Exploratory molecular biological investigations focusing on neurotrophic (e.g., BDNF, VEGF, GDNF) and immunological (e.g., TNF-alpha, IL-6, t-PA, S100A10) factors.
Epigenetic changes of neurotrophic and immunological factors at 4-week follow-up | From enrollment to 4 weeks after the end of iTBS treatment
  Exploratory molecular biological investigations focusing on neurotrophic (e.g., BDNF, VEGF, GDNF) and immunological (e.g., TNF-alpha, IL-6, t-PA, S100A10) factors.
Concentrations of markers of neuronal damage | From enrollment to the end of iTBS treatment
  Concentrations of markers of neuronal damage (e.g., NSE, S100-β) in serum.
Concentrations of markers of neuronal damage at 4-week follow-up | From enrollment to 4 weeks after the end of iTBS treatment
  Concentrations of markers of neuronal damage (e.g., NSE, S100-β) in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Schülke, MD (Dr. med.), Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Whether IPD may be shared has not yet been decided. IPD might not be shared due to data protection laws.